CLINICAL TRIAL: NCT04578600
Title: A Phase I/IB Pilot Study of CC-486 Combined With Lenalidomide and Obinutuzumab for Relapsed/Refractory Indolent B-Cell Lymphoma
Brief Title: CC-486, Lenalidomide, and Obinutuzumab for the Treatment of Recurrent or Refractory CD20 Positive B-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joseph Tuscano (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Celgene (Industry)
Responsible Party: Sponsor-Investigator, Joseph Tuscano, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1548998; NCI-2020-05946 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#282 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2020-09-21; First posted 2020-10-08 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Indolent B-Cell Non-Hodgkin Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Mucosa-Associated Lymphoid Tissue Lymphoma; Recurrent Follicular Lymphoma; Recurrent Hairy Cell Leukemia; Recurrent Lymphoplasmacytic Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Mucosa-Associated Lymphoid Tissue Lymphoma; Refractory Follicular Lymphoma; Refractory Hairy Cell Leukemia; Refractory Lymphoplasmacytic Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Leukemia, Hairy Cell; Lymphoma, Mantle-Cell | interventions — Lenalidomide; obinutuzumab; Azacitidine; cc-486

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (lenalidomide, oral azacitidine, obinutuzumab) (Experimental): Patients receive azacitidine PO QD on days 1-21, obinutuzumab IV over on days 8, 15, 22, and 29, and lenalidomide PO QD on days 8-28 of cycle 1. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity. Patients then receive azacitidine PO QD on days 1-21, obinutuzumab IV over on day 1, and lenalidomide PO QD on days 1-21. Cycles repeats every 28 days in the absence of disease progression, unacceptable toxicity, or until stem cell transplant. Patients who achieve SD, PR, or CR do not proceed to stem cell transplant may continue treatment for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide; Biological: Obinutuzumab; Drug: Oral Azacitidine

INTERVENTIONS:
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759
Drug: Oral Azacitidine — Given PO
  Other Names: CC-486

SUMMARY:
This phase I/Ib trial investigates the side effects of CC-486 and how well it works in combination with lenalidomide and obinutuzumab in treating patients with CD20 positive B-cell lymphoma that has come back (recurrent) or has not responded to treatment (refractory). Chemotherapy drugs, such as CC-486, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Lenalidomide is a drug that alters the immune system and may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may reduce or prevent the growth of cancer cells. Obinutuzumab is a type of antibody therapy that targets and attaches to the CD20 proteins found on follicular lymphoma cells as well as some healthy blood cells. Once attached to the CD20 protein the obinutuzumab is thought to work in different ways, including by helping the immune system destroy the cancer cells and by destroying the cancer cells directly. Giving CC-486 with lenalidomide and obinutuzumab may improve response rates, quality, and duration, and minimize adverse events in patients with B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To assess the safety and toxicity of oral azacitidine (CC-486) in combination with lenalidomide and obinutuzumab.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of CC-486 in combination with lenalidomide and obinutuzumab in subjects with relapsed/refractory indolent B-cell lymphoma as assessed by:

Ia. Overall response rate: complete response (CR) + partial response (PR) per 2016 Lugano criteria and Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC) criteria.

Ib. Duration of response (DOR): will be calculated from time of initial response assessment demonstrating at least PR until disease response assessment that demonstrates progressive disease.

Ic. Time to response (TTR): calculated as time from registration to first disease response assessment that demonstrates at least PR.

Id. Progression-free survival (PFS): Patients are considered a failure for this endpoint if they die or if they relapse/progress or receive additional anti-lymphoma therapy.

Ie. Determine the recommended phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* Previously treated, histologically confirmed CD20+ B cell lymphoma which includes mantle cell lymphoma, follicular lymphoma, chronic lymphocytic leukemia/small lymphocytic lymphoma, hairy cell leukemia, marginal zone lymphoma, mucosa-associated lymphoid tissue (MALT) lymphoma, and lymphoplasmacytic lymphoma. Fine needle aspirates are not acceptable
* Ability to understand and willingness to sign an informed consent form
* Ability to adhere to the study visit schedule and other protocol requirements
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1, or Karnofsky performance status (KPS) performance status of 60% or greater
* Life expectancy >= 3 months
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,000/uL
* Platelets >= 50,000/uL
* Total bilirubin: =< 2.0 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Serum creatinine

  * =< 2.0 x ULN, OR
  * Calculated creatinine clearance >= 30 ml/min/1.73 M^2 by the modified Cockcroft and Gault Formula, OR
  * Creatinine clearance >= 30 mL/min obtained from a 24-hour urine collection
* At least one measurable lesion according to International workshop lymphoma response criteria. There must be measurable lymphadenopathy to follow with serial exam and/or imaging
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study
* Submission of original biopsy for review and verification by participating center hematopathologist
* Disease free of prior malignancies for >= 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
* All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategies (REMS) program, and be willing and able to comply with the requirements of the REMS program
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation. (Subjects intolerant to acetylsalicylic acid [ASA] may use low molecular weight heparin)
* Must be able to swallow study drugs
* Human immunodeficiency virus (HIV) infected patients are eligible provided they meet all the other eligibility criteria of the study in addition to the following:

  * No history of acquired immunodeficiency syndrome (AIDS)-defining conditions other than lymphoma or history of CD4+ T-cells below 200/mm^3 prior to beginning combination antiretroviral therapy (cART)
  * After HIV diagnosis and during treatment with cART, patients should have maintained CD4+ T-cells >= 350/mm^3 prior to lymphoma diagnosis. Patents who never immune reconstituted to a stable level above 350/mm^3 are not eligible
  * At time of study entry CD4+ T-cells must have recovered from prior lymphoma therapy to >= 250/mm^3
  * At the time of study entry the HIV viral load must be undetectable by standard laboratory assay
  * During prior lymphoma therapy, patients must not have experienced documented infections attributed to the HIV+ status
  * No history of non-adherence to cART and willing to adhere to cART while on study
  * Antiretroviral drugs with overlapping or similar toxicity profiles as study agents not allowed:

    * Efavirenz not allowed due to potential central nervous system (CNS) toxicity
    * Stavudine not allowed due to potential neuropathic effects
    * Zidovudine not allowed due to myelosuppressive effects
  * Patients must be willing to be followed at a minimum of approximately every 3 months by physician expert in HIV disease management

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy within 28 days of baseline
* Known hypersensitivity to lenalidomide, thalidomide, obinutuzumab, or mannitol
* A history of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Any prior use of obinutuzumab or CC-486
* Concurrent use of other anti-cancer agents or treatments
* Known active hepatitis B or C. Patients on suppressive therapy with a negative viral load and no evidence of hepatic damage are eligible
* Uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment)
* Active central nervous system (CNS) involvement by lymphoma, including leptomeningeal involvement
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. A history of hemolytic anemia associated with the lymphoma does not exclude a patient from the study
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking azacitidine)
* For CC-486: History of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), celiac disease (i.e., sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the study drug (CC-486) and/or predispose the subject to an increased risk of gastrointestinal toxicity
* Abnormal coagulation parameters (prothrombin time [PT] > 15 seconds, partial thromboplastin time [PTT] > 40 seconds, and/or international normalized ratio [INR] > 1.5)
* Significant active cardiac disease within the previous 6 months including:

  * New York Heart Association (NYHA) class 4 congestive heart failure (CHF)
  * Unstable angina
  * Myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days post-last dose
  Safety summaries will include tabulations in the form of tables and listings. The frequency (number and percentage) of treatment-emergent AEs will be reported. The frequency of treatment-emergent AEs requiring discontinuation of study drug or dose reductions will be reported. Additional AE summaries will include AE frequency by AE severity and by relationship to study drug. Toxicity data by type and severity will be summarized by frequency tables. Per-treated analysis will be performed to include any patient who received the treatment regardless of the eligibility nor the duration or dose of the treatment received.

SECONDARY OUTCOMES:
Complete response rate | At 48 weeks
  Response will be assessed based on Cheson, Lugano classification 2016. The number and percentage of subjects with a complete response at 120 weeks will be tabulated.
Overall response rate (ORR) (complete response + partial response) | Up to 2 years
  Will be assessed by the investigator based on Cheson, Lugano classification 2016. The number and percentage of subjects with an ORR will be tabulated. The best ORR will be recorded.
Duration of response | From the time by which measurement criteria for complete response or partial response, whichever is recorded first, is met until death or the first date by which progressive disease is documented, assessed up to 2 years
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% confidence interval. Comparison by important subgroups will be made using the log-rank test.
Time to response | From registration to first disease response assessment that demonstrates at least partial response, assessed up to 2 years
  Comparison by important subgroups will be made using the log-rank test. Will be estimated using the product-limit method of Kaplan and Meier.
Progression-free survival | From the date of first dose (cycle 1, day 1) to the date of first documented progression or death, assessed up to 2 years.
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% confidence interval. Comparison by important subgroups will be made using the log-rank test.
Recommended phase 2 dose | Up to 35 days
  The maximum tolerated dose (MTD) will be defined as the highest dose of CC-486 tested in which fewer than 33% of patients experience a dose-limiting toxicity and at least 6 patients have been treated at that dose. The MTD will be the recommended phase 2 dose, provided that other safety considerations are acceptable.
Time to next treatment | From the end of cycle 24 (each cycle is 28 days) to the date of first documented new anti-lymphoma treatment, assessed up to 2 years.
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% confidence interval. Comparison by important subgroups will be made using the log-rank test.
Event-free survival | From the date of first dose (cycle 1, day 1) to the date of first documented progression, transformation to diffuse large B-cell lymphoma, initiation of new anti-lymphoma treatment, or death, assessed up to 2 years.
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% confidence interval. Comparison by important subgroups will be made using the log-rank test.
Overall survival | From the date of first dose (cycle 1, day 1) to the date of death regardless of cause, assessed up to years.
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% confidence interval. Comparison by important subgroups will be made using the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Tuscano, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States